CLINICAL TRIAL: NCT02977130
Title: The Influence of Conversation Map on the Health Behaviors of Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201404062RINB
Record Dates: First submitted 2016-11-24; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus; Health Knowledge, Attitudes, Practice; Health Behavior; Glycated Hemoglobin (HbA1c)
MeSH Terms: conditions — Diabetes Mellitus; Behavior; Health Behavior | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Map group (Experimental): patients receiving general shared care for diabetes and the conversation map intervention
  Interventions: Behavioral: Map group
- Control group (Active Comparator): patients receiving general shared care for diabetes
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Map group — diabetes shared care plus conversation map intervention
  Arms: Map group
Behavioral: Control group — diabetes shared care
  Arms: Control group

SUMMARY:
The American Diabetes Association indicates that diabetes self-management is a skill that diabetic patients must learn in the Diabetes Self-Management Education; thus, this contributes to shared care for diabetes, in which teams of physicians, professional nurses, and dietitians offer shared care to patients. However, according to the statistical analysis of the conditions of glycemic control in diabetic patients in 28 countries across 4 continents (Asia, Africa, Europe, and South America), the mean glycated hemoglobin (HbA1c) of the 12,727 patients was 9.5% by Litwak et al. in 2013. In Taiwan, a national survey among diabetic patients in a shared-care program found that the percentage of patients with HbA1c lower than 7% increased by 6.5% from 2006 to 2011; yet, among the 720 patients who completed both surveys in 2006 and 2011, the percentage with HbA1c lower than 7% decreased by 2.1% during that period. These results suggest that despite the increase in the proportion of patients who successfully managed their diabetes, some patients still encountered difficulty in glycemic control.Therefore, numerous health education tools on diabetes continue to be developed. In 2011,JoAnn et al. determined that the mode of health care had a substantial influence on the dietary habits of diabetic patients, and that individual health education had the largest effect on diabetes control. In addition, using the conversation map for diabetes control also had a substantial influence on improving health behaviors. Among existing studies that have adopted the conversation map, no large-scale research has been conducted, the research samples and relevant studies in Taiwan have been scant, and no theoretical foundation has been applied in evaluating the effects of the conversation map. Accordingly, the investigators aimed to enhance the mutual experience exchange and learning among diabetic patients through adopting the conversation map to observe its influence on their health behaviors by incorporating it into existing health education modalities. Furthermore, on the basis of the Health Belief Model, a relevant questionnaire was designed for assessing the effectiveness of glycemic control in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus between 30 and 80 years of age who participated in a diabetes shared-care program.

Exclusion Criteria:

* Patients were excluded if they had renal insufficiency (eGFR <30 mL•min / 1.732), were not ambulatory, or were unable to answer the questionnaire independently.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Diet- and exercise-related health behaviors | 3 months
Glycated hemoglobin (HbA1c) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jiun-Hau Huang, SM, ScD, Principal Investigator — National Taiwan University

IPD SHARING:
Plan to Share IPD: No